CLINICAL TRIAL: NCT05732220
Title: Mobile Ecological Momentary Assessment-based Peer Counselling for Youth Smokers: a Pilot Randomised Controlled Trial
Brief Title: Mobile EMA-based Peer Counselling for Youth Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tzu Tsun Luk, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202111159206
Record Dates: First submitted 2023-02-05; First posted 2023-02-16 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation
Keywords: counselling; ecological momentary assessment; young smoker; mobile health; adolescsent; quitline; Chinese
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EMA+ group (Experimental): EMA assessment + EMA-based cessation counselling
  Interventions: Behavioral: EMA assessment; Behavioral: EMA-based cessation counselling
- EMA group (Active Comparator): EMA assessment only + Usual peer counselling
  Interventions: Behavioral: EMA assessment; Behavioral: Usual peer counselling
- Control (Active Comparator): Usual peer counselling
  Interventions: Behavioral: Usual peer counselling

INTERVENTIONS:
Behavioral: EMA assessment — Subjects will be asked to complete 3 waves of ecological momentary assessment (EMA) about smoking cues and smoking consumption via mobile phone at the first, second and third month after baseline (total 6 weeks)
  Arms: EMA group; EMA+ group
Behavioral: EMA-based cessation counselling — Subjects will receive tailored peer counselling based on the participants' EMA responses at 1-month and 3-month telephone follow-ups.
  Arms: EMA+ group
Behavioral: Usual peer counselling — Subjects will receive peer counselling through telephone during follow-ups (usual care), in which the counsellor will apply the 5As model and motivational interviewing techniques.
  Arms: Control; EMA group

SUMMARY:
This pilot trial aims to examine the feasibility, acceptability, and preliminary effectiveness of EMA-based peer counseling for youth smokers.

DETAILED DESCRIPTION:
Most smokers begin smoking during adolescence and early adulthood, a crucial period to prevent initiation and continuation of smoking. However, many proven smoking cessation interventions for adult smokers were not found effective in youth smokers, which may be partly explained by the vast differences in the pattern of tobacco use and determinants of quitting between adult and youth smokers. This calls for more research on novel intervention models to help young smokers quit.

The HKU Youth Quitline provides free smoking cessation support for smokers aged below 25 years since August 2005 in Hong Kong. The service provides multisession peer-led telephone counselling with an individualised quit plan devised for each young smoker according to their responses. Since the counselling model depends on the information retrospectively recalled by the smokers, it may be prone to recall and social desirability biases and fail to capture the variability of youth smoking patterns and momentary changes in personal (e.g., mood) and situational (e.g., peer smoking) antecedents of smoking episodes.

Recent advances in mobile technologies have enabled the use of more advanced and robust data collection approaches like ecological momentary assessment (EMA), which may benefit the counselling model by providing more ecologically valid data than traditional surveys. Previous studies have demonstrated the feasibility of using EMA to collect data on psychosocial processes and smoking behaviours in adolescent smokers. Therefore, we propose to develop and test a mobile EMA-based counselling intervention for youth smokers by conducting a pilot RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15 to 25 years
2. Have smoked in the past 30 days
3. Own a smartphone with an mobile instant messaging app installed
4. Can communicate in Chinese

Exclusion Criteria:

Youth smokers who are participating in other smoking cessation studies or program other than the HKU Youth Quitline

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically-validated tobacco abstinence | 6 months after randomisation
  Defined as a negative result of the iScreen OFD test for measuring salivary cotinine (with a cut-off of lower than 30ng/mL)

SECONDARY OUTCOMES:
Self-reported 7-day point-prevalence tobacco abstinence | 3 months after randomisation
  Being completely smoke-free in the past 7 days
Self-reported 7-day point-prevalence tobacco abstinence | 6 months after randomisation
  Being completely smoke-free in the past 7 days
Self-reported 30-day point-prevalence tobacco abstinence | 3 months after randomisation
  Being completely smoke-free in the past 30 days
Self-reported 30-day point-prevalence tobacco abstinence | 6 months after randomisation
  Being completely smoke-free in the past 30 days
Smoking reduction by at least 50% | 3 months after randomisation
  Smoking reduction by at least half of the baseline daily number of cigarettes
Smoking reduction by at least 50% | 6 months after randomisation
  Smoking reduction by at least half of the baseline daily number of cigarettes

OTHER OUTCOMES:
Recruitment rate | Through recruitment completion, about 6 months
  Proportion of participants among all eligible subjects
Retention rate | 6 months after randomisation
  Proportion of participants responding to telephone follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Tsun Luk, PhD, RN, Principal Investigator — The University of Hong Kong
Locations (1):
- HKU Youth Quitline, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan SS, Wong DC, Fong DY, Leung AY, Lam DO, Mak YW, Lam TH. The establishment and promotion of the first Youth Quitline in Hong Kong: challenges and opportunities. Eval Health Prof. 2008 Sep;31(3):258-71. doi: 10.1177/0163278708320156. Epub 2008 Jun 19. PMID 18566161
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Van Zundert RM, Ferguson SG, Shiffman S, Engels R. Dynamic effects of craving and negative affect on adolescent smoking relapse. Health Psychol. 2012 Mar;31(2):226-34. doi: 10.1037/a0025204. Epub 2011 Sep 26. PMID 21942749
- [Background] McClure EA, Tomko RL, Carpenter MJ, Treiber FA, Gray KM. Acceptability and compliance with a remote monitoring system to track smoking and abstinence among young smokers. Am J Drug Alcohol Abuse. 2018;44(5):561-570. doi: 10.1080/00952990.2018.1467431. Epub 2018 May 8. PMID 29737885
- [Background] Fanshawe TR, Halliwell W, Lindson N, Aveyard P, Livingstone-Banks J, Hartmann-Boyce J. Tobacco cessation interventions for young people. Cochrane Database Syst Rev. 2017 Nov 17;11(11):CD003289. doi: 10.1002/14651858.CD003289.pub6. PMID 29148565